CLINICAL TRIAL: NCT05352126
Title: Effects of Repeated Sprays of an Air Purifying Spray Containing Essential Oils in an Indoor Environment on Asthma Control in Patients With Mild to Moderate Allergy-induced Asthma.
Brief Title: Effects of Puressentiel Purifying Spray on Asthma Control in Patients With Mild to Moderate Allergy-induced Asthma.
Acronym: PSIndAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Puressentiel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Prof. Pascal Demoly
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Asthma, Allergic
MeSH Terms: conditions — Asthma | interventions — Disinfectants

STUDY DESIGN:
Intervention Model Description: Multicentre prospective cross-over, randomised, double-blind placebo-controlled trial
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puressentiel Purifying spray (Experimental): Puressentiel Air Purifying Spray with 41 essential oils
  Capacity: 200 ml
  BIOCIDE Product type 2: Disinfectants used in the private and public health sector
  Composition: Ethanol (CAS no. 64-17-5) 75% m/m and 41 essential oils
  Interventions: Other: Biocide
- Placebo (Placebo Comparator): Saline spray in the similar device as Puressentiel Purifying spray
  Interventions: Other: Biocide

INTERVENTIONS:
Other: Biocide — The product being researched, which is a biocide solution in a spray for atmospheric use without a propellant, will be sprayed in the bedroom of each patient at a rate of 2 sprays per day in the evening (half an hour before going to bed).

SUMMARY:
The main objective of this study is to evaluate, in real life, the efficacy of prolonged use (6 months) of Puressentiel Air Purifying Spray with 41 essential oils on the control of allergy-induced asthma in the homes of patients with mild to moderate asthma. This will be performed by evaluating the efficacy of prolonged use (6 months) in the indoor environment on the exacerbation and the symptoms of asthma in patients with mild to moderate asthma. The tolerance of the study patients to spraying in an indoor environment will also be analysed.

DETAILED DESCRIPTION:
At the inclusion visit (V1), the number of exacerbations requiring oral corticosteroids, and asthma treatments (base and rescue medication) during the previous 12 months are collected.

An Asthma Control Test (ACT) for self-assessment is given to the patient. This questionnaire (Appendix 1) contains 5 questions related to asthma symptoms and their frequency as well as the rescue medication used in the previous 4 weeks. The ACT score ranges from 5 (most badly controlled) to 25 (fully controlled asthma). The threshold for controlled asthma is 20, with a lower score indicating uncontrolled asthma. (14).

Vials of Puressentiel Air Purifying Spray with 41 essential oils or weighed identical placebo bottles are given to the patient according to the randomisation period that he/she has been assigned to. The patient is asked to spray in 2 corners of the bedroom (at bedtime (2/D) for 6 months). A telephone visit will be carried out by the CRA of the study at 3 months (see telephone visit). At the end of the 6 months, the subject is reviewed (V2) and will bring back the used spray bottles which will be weighed to assess compliance. In a second Asthma Control Test (ACT), the number of exacerbations, during the 6 months of use of Puressentiel Air Purifying Spray with 41 essential oils or the placebo is collected. Bottles of placebo air spray or Puressentiel Air Purifying Spray with 41 essential oils are given to the patient according to the randomisation period that he/she has been assigned to during the first visit (V1).

The patient is seen again 6 months later (V3), during which time he/she will use the placebo spray or Puressentiel Air Purifier Spray with 41 essential oils, one spray in 2 corners of the bedroom (i.e. 2 sprays in total) in the evening (2/D). A second Asthma Control Test (ACT) is performed and the number of exacerbations over the 6 months is collected. A telephone visit will be carried out by the CRA of the study at 9 months (see telephone visit).

If the patient has been randomised to receive the placebo spray during the first six-month period, he/she will use Puressentiel Air Purifying Spray with 41 essential oils during the second six-month period.

ELIGIBILITY:
Inclusion Criteria:

* • Mild to moderate asthma patients with or without rhinitis who were diagnosed with asthma at least one year beforehand. At least partially controlled (16≥ACT≥23)

  * Patients who are allergic to one allergen per year and/or season (proof of prick tests or specific IgE).
  * Patients who are over 18 years old.
  * Patients who have read and signed the informed consent form
  * Patients who are affiliated to the social security regime

Exclusion Criteria:

* • Patients who have had a viral infection in the month prior to inclusion

  * Patients with uncontrolled asthma.
  * Pregnant or breastfeeding women.
  * People with a history of seizure disorders, or epilepsy
  * People with allergies to any of the components of the product
  * Patients with comprehension difficulties
  * Patients who cannot be monitored throughout the entire period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Asthma control | 6 months
  The primary endpoint of this study is the Asthma Control Test (ACT), which is assessed after 6 months of exposure and compared to 6 months without exposure, with the patient being his or her own control. A difference of 2 points questionnaire ranging from 5 to 25 is considered clinically significant

SECONDARY OUTCOMES:
Exacerbation of asthma | 6 months
  Number of exacerbations

IPD SHARING:
Plan to Share IPD: No